CLINICAL TRIAL: NCT04778384
Title: Evaluation of the Effectiveness of a Patient Education for Oncological Patients to Promote Self-management in Pain Therapy
Brief Title: Patient Education to Promote Self-management in Pain Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intervention_Pain_Therapy
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-04

CONDITIONS: Patient Empowerment
MeSH Terms: conditions — Patient Participation | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: Data analysis with statistical process control:
  Data is collected in two time series. First, data of patients with sham intervention (control intervention) is collected, then data is collected from patients with a structured micro-training (study intervention).
Who Masked: Participant
Masking Description: Patients do not know which training series they belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 30 patients receive micro-training based on a checklist & targeted discussion / dismantling of patient-related barriers based on the answers in the second part of the questionnaire (BQII Barriers Questionnaire)
  Interventions: Behavioral: Micro-training to promote self-management in pain therapy
- Control Group (Sham Comparator): 30 patients receive a sham intervention: an unstructured conversation is carried out. Patient questions are answered correctly, but there is no training, rather patient information.
  Interventions: Other: Sham intervention

INTERVENTIONS:
Behavioral: Micro-training to promote self-management in pain therapy — Micro-training according to the checklist & targeted discussion / dismantling of patient-related barriers based on the answers in the second part of the questionnaire (BQII Barriers Questionnaire) In this discussion, the nurses give their opinion on any patient-related barriers that become apparent after completing the second part of the questionnaire. This is not done according to a fixed template, but with the specialist knowledge and everyday experience of the nurse.
  Arms: Intervention Group
Other: Sham intervention — An unstructured conversation is carried out. Patient questions are answered correctly, but there is no training, rather patient information.
  Arms: Control Group

SUMMARY:
Monocentric, uncontrolled before / after study to evaluate the effectiveness of a patient education for oncological patients by nursing staff to promote self-management in pain therapy.

The structured patient education (in the form of a micro-training) is intended to specifically promote pain self-management in oncological patients. In contrast to conventional training courses, this requires the patient to be actively involved in the process so that the skills learned can be used to optimally adapt the therapy on an individual level. Through the intervention, we postulate the advantage that the increased self-management of pain therapy improves the everyday functions of the patient, and by breaking down patient-related barriers and checking the accessibility of pain medication, the safety in dealing with pain therapy and thus patient satisfaction increases.

Data is collected in two time series. First, data of patients with sham intervention (control intervention) is collected, then data is collected from patients with a structured micro-training (study intervention). Patients do not know which training series they belong to.

DETAILED DESCRIPTION:
Nursing staff is trained to conduct the micro-training. The sham intervention is unstructured at the discretion of the respective nurse. They are only informed about the purpose of the sham intervention, the expected time frame and the course of a sample sham intervention.

First, the data collection of the group with control intervention is started until the required number of patients is recorded. As soon as these data are complete, the group with study intervention is recorded.

The patients are recruited from the oncological outpatient clinics. After the outpatient clinics before a parenteral therapy, they have a waiting period, during which the patient's consent is obtained. The patients are then taken to the intervention room for parenteral therapy. Here, the questionnaire is filled out before, during or after the therapy, and then the intervention with the nurse takes place. This process with a short reflection period must be designed in such a way because the indication for escalation of the opioid pain treatment is made during the oncological consultation which is the only possibility to recruit patients for this pilot study. The way the clinic runs today, the nursing staff is timewise only available for training patients with parenteral therapy. If the patients needed more time to think about it, they would have to be trained separately at a later point in time, which would only be established if the effectiveness of the patient training could be proven. Because the patients are not exposed to any risk from the planned interventions, this procedure is reasonable in our view.

In micro-training (study intervention), patients are taught structured knowledge based on the content of a checklist. In addition to pain recording, patients are trained in the use of basic and reserve pain medication and co-analgesics, the most common opioid side effects are discussed and how to react to them. It is also checked that the necessary prescriptions or medication have been given. Furthermore, after completing the BQII Barriers Questionnaire (second part of the questionnaire), patient-related barriers, i.e. concerns or fears of the patient with regard to pain therapy, become apparent. With a factual discussion and a professional weighing of advantages and disadvantages, the nurse tries to break down these barriers and thus promotes the patient's motivation for a well-adapted pain therapy. In the case of sham intervention (control intervention), there is only a conversation between the nurse and the patient. In this conversation the patient is picked up with his current knowledge about his pain therapy and any questions are answered correctly. However, there is no structured transfer of knowledge in the sense of patient training.

The data is recorded using a three-part questionnaire. The first part of the questionnaire contains questions regarding pain-related restrictions in everyday activities (using the Brief Pain Inventory as the standard for pain assessment of oncological patients as used by the Swiss Cancer League). The second part of the questionnaire deals with patient-related barriers using the BQII Barriers Questionnaire. The third part of the questionnaire consists of global questions: confidence in dealing with pain medication, satisfaction with pain therapy, restriction of the most important activities in everyday life and satisfaction with quality of life.

4 weeks after the intervention, patients are asked to fill in the same three-part questionnaire again. At that time, the questionnaire is sent to them by mail with a reply envelope.

ELIGIBILITY:
Inclusion Criteria:

• Oncology clinics outpatients with parenteral therapy with a new or escalated opioid pain therapy without exclusion criteria

Exclusion Criteria:

* Lack of consent
* Insufficient knowledge of German
* Cognitive deficits

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain-related restriction of daily activities | 20 months
  Questionnaire part 1: according to the Brief Pain Inventory Scale title: Do you feel restricted in everyday life because of the pain? 8 items with possible answers on a 5-pt-Likert-scale ranging from "not restricted" = 1pt to "completely restricted" = 5pts minimum score 8pts, maximum score 40pts with higher scores meaning a worse outcome

SECONDARY OUTCOMES:
Change in patient-related barriers | 20 months
  Questionnaire part 2: according to the BQII Barriers Questionnaire Scale title: We are interested in your attitude towards pain therapy. Please tick the box that most applies to you.
  12 items with possible answers on a 5-pt-Likert-scale ranging from "completely disagree" = 1pt to "completely agree" = 5pts possible minimum score 12pts, possible maximum score 60pts with higher scores meaning a worse outcome (meaning higher barriers towards pain therapy)
Confidence in handling pain medication, satisfaction with pain therapy and quality of life, restriction of the most important activities in everyday life | 20 months
  Questionnaire part 3: recorded with global questionsScale title: Please tick the box that most applies to you.
  4 global questions regarding self competence and satisfaction with pain therapy, the ability to fulfill the most important daily activity despite the pain and overall satisfaction with quality of life.
  Possible answers on a 5-pt-Likert-scale ranging from "completely disagree" = 1pt to "completely agree" = 5pts possible minimum score 4pts, possible maximum score 20pts with higher scores meaning a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Fabia Buettcher, MD, Study Chair — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raphaelis S, Frommlet F, Mayer H, Koller A. Implementation of a nurse-led self-management support intervention for patients with cancer-related pain: a cluster randomized phase-IV study with a stepped wedge design (EvANtiPain). BMC Cancer. 2020 Jun 16;20(1):559. doi: 10.1186/s12885-020-06729-0. PMID 32546177